CLINICAL TRIAL: NCT00828061
Title: A Randomized Clinical Trial to Study the Effects of Single Dose of Corticosteroid on Response to Nasal Allergen Challenge in Patients
Brief Title: A Study of the Effects of Single Dose Corticosteroids on Response to Allergens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-129; 2009_517
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Results first posted 2010-05-05 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- B (Active Comparator): 10 mg prednisone
  Interventions: Drug: prednisone
- C (Active Comparator): 25 mg prednisone
  Interventions: Drug: prednisone

INTERVENTIONS:
Drug: Placebo — Single dose of 5 tablets matching placebo (5 x 0 mg) to prednisone. The washout between treatment periods will be approximately 4 weeks
  Arms: A
Drug: prednisone — Single dose of 5 tablets prednisone totaling 10 mg (3 x 0 mg + 2 x 5 mg). The washout between treatment periods will be approximately 4 weeks.
  Arms: B
Drug: prednisone — Single dose of 5 tablets prednisone totaling 25 mg (5 x 5 mg). The washout between treatment periods will be approximately 4 weeks.
  Arms: C

SUMMARY:
This study will investigate whether changes in inflammatory mediators produced by the nose after exposure to an allergen can be used to evaluate the anti-inflammatory effects of novel drugs for the treatment of allergic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patient is allergic to Timothy grass pollen
* Female patients have a negative pregnancy test and agree to use birth control throughout the study
* Male patients agree to use birth control throughout the study
* Patient has been a nonsmoker for at least 6 months
* Patient agrees to avoid the use of aspirin and other Non-steroidal anti-inflammatory drugs (NSAIDs) throughout study

Exclusion Criteria:

* Patient is breastfeeding
* Patient has any respiratory disease other than mild stable asthma that does not require treatment
* Patient consumes more than 3 alcoholic beverages per day
* Patient consumes more than 6 caffeinated beverages per day
* Patient has had major surgery or has donated or lost 1 unit of blood within 4 weeks of screening
* Patient has severe allergies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-02-04 (Actual); Primary Completion 2009-05-07 (Actual); Study Completion 2009-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Leaker BR, Malkov VA, Mogg R, Ruddy MK, Nicholson GC, Tan AJ, Tribouley C, Chen G, De Lepeleire I, Calder NA, Chung H, Lavender P, Carayannopoulos LN, Hansel TT. The nasal mucosal late allergic reaction to grass pollen involves type 2 inflammation (IL-5 and IL-13), the inflammasome (IL-1beta), and complement. Mucosal Immunol. 2017 Mar;10(2):408-420. doi: 10.1038/mi.2016.74. Epub 2016 Sep 28. PMID 27677865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Entered: 04-Feb-2009
  Last Patient, Last Visit: 21-May-2009
  2 sites
Groups:
- Placebo / Prednisone / Prednisone: 1 day placebo, 1 day 10 mg prednisone, 1 day 25 mg prednisone
- Prednisone / Prednisone / Placebo: 1 day 10 mg prednisone, 1 day 25 mg prednisone, 1 day placebo
- Prednisone / Placebo / Prednisone: 1 day 25 mg prednisone, 1 day placebo, 1 day 10 mg prednisone
- Placebo / Prednisone / Prednisone: 1 day placebo, 1 day 25 mg prednisone, 1 day 10 mg prednisone
- Prednisone / Placebo / Prednisone: 1 day 10 mg prednisone, 1 day placebo, 1 day 25 mg prednisone
- Prednisone / Prednisone / Placebo: 1 day 25 mg prednisone, 1 day 10 mg prednisone, 1 day placebo
Period: Period 1
Arm/Group | Placebo / Prednisone / Prednisone | Prednisone / Prednisone / Placebo | Prednisone / Placebo / Prednisone | Placebo / Prednisone / Prednisone | Prednisone / Placebo / Prednisone | Prednisone / Prednisone / Placebo
Started | 4 | 3 | 3 | 3 | 3 | 3
Completed | 4 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Placebo / Prednisone / Prednisone | Prednisone / Prednisone / Placebo | Prednisone / Placebo / Prednisone | Placebo / Prednisone / Prednisone | Prednisone / Placebo / Prednisone | Prednisone / Prednisone / Placebo
Started | 4 | 3 | 3 | 3 | 3 | 3
Completed | 4 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Placebo / Prednisone / Prednisone | Prednisone / Prednisone / Placebo | Prednisone / Placebo / Prednisone | Placebo / Prednisone / Prednisone | Prednisone / Placebo / Prednisone | Prednisone / Prednisone / Placebo
Started | 4 | 3 | 3 | 3 | 3 | 3
Completed | 4 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: All patients who completed at least one period are included in the analysis
Arm/Group | All Patients
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 40.4 [22 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Fold Change From Baseline at Hour 8 in Interleukin 5 (IL-5) Concentration
Description: Comparison of the Change in Allergen-induced Interleukin 5 (IL-5) as Measured in Nasal Exudates After a Single Dose of Low or High Dose of Oral Prednisone Relative to Placebo
Time Frame: Baseline and Hour 8 post nasal allergen challenge
Population: All Patients as Treated
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Placebo | 10 mg Prednisone | 25 mg Prednisone
Number analyzed (Participants) | 19 | 19 | 19
Fold Change | 26.94 [7.33 to 99.00] | 6.70 [1.82 to 24.61] | 1.86 [0.51 to 6.83]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Prednisone; Test type: Superiority or Other; p = 0.002, ANOVA — 1-sided, alpha = 0.05; Analysis performed on log-transformed fold change from baseline and results were back-transformed for reporting; Geometric Mean Fold Difference = 0.25, 95% CI [0.12 to 0.54]
Statistical Analysis 2: Comparison: Placebo vs 25 mg Prednisone; Test type: Superiority or Other; p < 0.001, ANOVA — 1-sided, alpha = 0.05; Analysis performed on log-transformed fold change from baseline and results were back-transformed for reporting; Geometric Mean Fold Difference = 0.07, 95% CI [0.03 to 0.15]

2. Secondary Outcome: Change From Baseline at Hour 8 in the Percent of Total Cells That Are Eosinophils
Description: Comparison of the Change in the Percent of Total Cells That Are Eosinophils Measured in Nasal Lavage After a Single Dose of 10 mg or 25 mg Prednisone Relative to Placebo
Time Frame: Baseline and Hour 8 post nasal allergen challenge
Population: All Patients with Slide Quality ≤ 3 (Slide Quality measured on a 6 point scale with values > 3 indicating a level of debris that interferes with cell typing and counting).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of cells that are eosinophils
Arm/Group | Placebo | 10 mg Prednisone | 25 mg Prednisone
Number analyzed (Participants) | 6 | 8 | 9
Percentage of cells that are eosinophils | 2.28 [-12.33 to 16.79] | 3.17 [-9.19 to 15.52] | 6.02 [-4.17 to 16.21]
Statistical Analysis 1: Comparison: Placebo vs 10 mg Prednisone; Test type: Superiority or Other; p = 0.537, ANOVA — 1-sided, alpha = 0.05; Mean Difference (Final Values) = 0.89, 95% CI [-15.48 to 17.26]

ADVERSE EVENTS:
Time Frame: Adverse experiences were collected from the time the consent is signed through the 14 day follow up period after all treatment periods were completed.
Description: AE s were assessed by clinical evaluation including vital signs, physical examination, medical history, clinical laboratory safety assessment (hematology, chemistry, urinalysis), and Electrocardiogram (ECG) at timepoints specified in the study. Patients were queried at each visit for any adverse experiences since the previous visit.
Arm/Group | Placebo | 10 mg Prednisone | 25 mg Prednisone
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 12/19 | 8/19 | 8/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | 10 mg Prednisone (N=19) | 25 mg Prednisone (N=19)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Oral Herpes (Infections and infestations) | 1 | 2 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0 | 0
Culture Urine Positive (Investigations) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 2 | 0 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 1
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Rhinitis Seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper Airway Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Poor cell yields from nasal lavage significantly reduced the utility of eosinophil count data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.